CLINICAL TRIAL: NCT00194376
Title: Evaluation of Gastroesophageal Reflux in Patients on Continuous Positive Airway Pressure Ventilation for Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: David C. Metz, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 802805
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Gastroesophageal Reflux; Sleep Apnea
MeSH Terms: conditions — Gastroesophageal Reflux; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

INTERVENTIONS:
Procedure: Continuous positive airway pressure ventilation — CPAP ventilation is a therapeutic modality which uses positive pressure of air through a sealed nasal mask to treat a condition known as sleep apnea

SUMMARY:
Patients with a clinically indicated sleep study will be enrolled in this study. They will have a diagnostic and a therapeutic sleep study with continuous positive airway pressure ventilation. For both studies a pH probe will be placed nasal to measure the amount of acidic reflux during each study. Baseline levels of reflux from the diagnostic sleep study will be compared to reflux episodes while on continuous positive airway pressure ventilation.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age, symptoms consistent with sleep apnea, agree to consent form and placement of pH probes

Exclusion Criteria:

* any unstable medical condition, previous upper gi surgery or anatomic abnormality of upper gi tract, acid suppressing medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2005-06; Primary Completion 2006-09 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Decrease in GERD symptoms | 24 hours
  Patients suffering from Obstructive Sleep Apnea have been shown to suffer from GERD events more frequesntly and with prolonged episodes compared to controls.

CONTACTS AND LOCATIONS:
Overall Officials: David Metz, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States